CLINICAL TRIAL: NCT02733094
Title: Single-arm Study to Assess a Potential Effect of Anti-IL-17 (Secukinumab) in the Treatment of Pyoderma Gangrenosum
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN547ADE01T
Record Dates: First submitted 2016-03-28; First posted 2016-04-11 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2020-02

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label (Experimental): 300 mg secukinumab every week for 4 weeks followed by 300 mg secukinumab every 2 weeks until week 32.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab

SUMMARY:
The purpose of this study is to explore the efficacy and safety of anti-Interleukin-(IL)17 therapy (secukinumab, administered weekly for 4 weeks followed by four-weekly administration until week 16) for the treatment of pyoderma gangrenosum.

ELIGIBILITY:
* Key Inclusion Criteria:

  * Confirmed diagnosis of Pyoderma gangrenosum
  * Biopsy-proven, non-healing ulcer with primarily neutrophil infiltration, regardless of size and location
  * Characterization of target lesion (size, PGA, duration)
  * 18-75 years of age
  * Body weight ≥ 40 kg and ≤ 160 kg
  * Signed informed consent
* Key Exclusion Criteria:

  * Permanent severe diseases, especially those affecting the immune system
  * Pregnancy or breast feeding
  * History or presence of epilepsy, significant neurological disorders, cerebrovascular attacks or ischemia
  * Myocardial infarction or cardiac arrhythmia which requires drug therapy
  * Evidence of severe renal dysfunction or significant hepatic disease
  * History of irritable bowel disease
  * History of lymphoproliferative disorders
  * Evidence for active infection including but not limited to active tuberculosis, HIV or hepatitis B/C that in the opinion of the investigator would compromise the patient's ability to tolerate therapy
  * History of malignancy of any organ system, treated or untreated, whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04; Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Change of the Physician's global assessment | Week 16
  The primary response parameter change of the physician global assessment (PGA) 5-point scale at week 16 as compared to week 0.

SECONDARY OUTCOMES:
Change in surface area of lesions of pyoderma gangrenosum (two-dimensional surface in mm²) | Week 2,3,8,16,28,40
Assessment of patient's quality of life | Week 2, 4, 8, 16, 28, 40
  Patient's quality of life is assessed by the Dermatology Life Quality Index (DLQI) questionnaire.
Measurement of serum C reactive protein (mg/dl) | Week 2, 4, 8, 16, 28, 40
Measurement of leukocyte counts (x10.e3/µl) | Week 2, 4, 8, 16, 28, 40
Measurement of blood sedimentation rate (mm/h) | Week 2, 4, 8, 16, 28, 40
Immunohistochemical analysis of IL-17+ immune cells | Week 16
  The number of IL-17+ immune cells is counted in two high-power-fields (400x) and mean in calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Kilian Eyerich, MD, PhD, Principal Investigator — Technical University of Munich
Locations (1):
- Technical University of Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided